CLINICAL TRIAL: NCT01235936
Title: Phase 2a Open-Label Pilot Study to Assess the Pharmacodynamic Response, Pharmacokinetics, Safety, and Tolerability of 28-Day Repeat Oral Doses of AKB-6548 in Subjects With Anemia Secondary to Chronic Kidney Disease (CKD), Stages 3 and/or 4
Brief Title: Safety and Efficacy Study for AKB-6548 in Participants With Chronic Kidney Disease and Anemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Akebia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AKB-6548-CI-0004
Record Dates: First submitted 2010-11-05; First posted 2010-11-08 (Estimated); Results first posted 2022-07-01 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Anemia; Kidney Disease
Keywords: anemia; chronic kidney disease; CKD; chronic renal insufficiency; renal impairment; erythropoietin; safety; efficacy; tolerability; pharmacokinetics
MeSH Terms: conditions — Anemia; Kidney Diseases; Renal Insufficiency, Chronic; Renal Insufficiency | interventions — vadadustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AKB-6548 (Experimental)
  Interventions: Drug: AKB-6548

INTERVENTIONS:
Drug: AKB-6548 — Different dose levels

SUMMARY:
The purpose of this study is to evaluate the safety, pharmacodynamics and pharmacokinetics of repeat doses of orally administered AKB-6548 in pre-dialysis participants with anemia.

ELIGIBILITY:
Key Inclusion Criteria:

* 18 to 79 years of age, inclusive
* Chronic Kidney Disease Stage 3 or Stage 4
* Hemoglobin (Hgb) < 10.5 g/dl
* TSAT > 20% and CBC indicating normocytic red blood cell morphology

Key Exclusion Criteria:

* BMI > 40
* Red blood cell transfusion within 12 weeks.
* Androgen therapy within the previous 21 days prior to study dosing
* Therapy with any approved or experimental erythropoiesis stimulating agent (ESA) within the 10 weeks prior to the Screening visit
* Participants meeting the criteria of ESA resistance within the previous 4 months
* Individual doses of intravenous iron of 250 mg or larger within the past 21 days
* AST or ALT >1.8x ULN.
* Alkaline phosphatase >2x ULN.
* Total bilirubin >1.5x ULN.
* Uncontrolled hypertension
* New York Heart Association Class III or IV congestive heart failure
* Myocardial infarction, acute coronary syndrome, or stroke within 6 months prior to dosing

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-10-21; Primary Completion 2011-04-13 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Akebia Therapeutics Inc.
Locations (2):
- United States (2):
  - Augusta, Georgia
  - San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study enrolled Chronic Kidney Disease (CKD) Stage 3 or CKD Stage 4 participants. Per protocol, this is a pilot study and all results data are summarized as a single treatment arm (i.e., all participants receiving Vadadustat); no separate analysis was performed to report results by disease state as the Sponsor terminated the study early after enrolling 10 participants.
Groups:
- Vadadustat: Participants received Vadadustat orally, once daily for 28 days. Participants with Stage 3 and Stage 4 CKD started dosing with 400 milligrams (mg) and 300 mg Vadadustat, respectively. Thereafter, at each of the weekly study visits, dose adjustments were made based on pre-defined dose adjustment algorithm in 100 mg increments allowing a dose range of 200 mg/day to 700 mg/day for Stage 3 CKD participants and 200 mg/day to 600 mg/day for Stage 4 CKD participants.
Period: Overall Study
Arm/Group | Vadadustat
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: All participants who received at least 1 dose of study medication. Per the protocol, all results data are summarized as a single treatment arm (i.e., all participants receiving Vadadustat); no separate analysis was performed to report results by disease state.
Arm/Group | Vadadustat
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.1 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 4
  More than one race | 0
  Unknown or Not Reported | 1
Kidney disease stage [Count of Participants; unit: Participants] — Stage 3 CKD: estimated glomerular filtration rate (eGFR) of 30-59 millilitre/minute/1.73 meter square (mL/min/1.73m^2) (moderate kidney damage).
  Stage 4 CKD: eGFR of < 30 mL/min/1.73m^2; participant was not yet on dialysis and not expected to start dialysis within the next 3 months (severe kidney damage).
  Participants
    Stage 3 | 6
    Stage 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Hemoglobin (Hgb) on Day 29
Description: Blood samples were collected to assess Hgb. Baseline Hgb was defined as the average of the 2 samples obtained prior to dosing (Pre-Baseline and Baseline). A positive change from baseline indicates that hemoglobin concentration increased.
Time Frame: Baseline; Day 29
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Grams per decilitre (g/dL)
Arm/Group | Vadadustat
Number analyzed (Participants) | 10
Grams per decilitre (g/dL)
  Baseline | 9.91 (0.63)
  Change from Baseline on Day 29 | 0.63 (0.46)
Statistical Analysis 1: Comparison: Vadadustat; Analysis of change from baseline on Day 29; Test type: Other — The primary endpoint was compared using the Wilcoxon signed-rank test, with an alpha level of 0.05; p = 0.0020, Wilcoxon signed rank test

2. Secondary Outcome: Mean Change From Baseline in Hematocrit on Day 29
Description: Blood samples were collected to assess hematocrit. A positive change from baseline indicates hematocrit concentration increased.
Time Frame: Baseline; Day 29
Population: Full analysis set population. Per the protocol, all results data are summarized as a single treatment arm (i.e., all participants receiving Vadadustat); no separate analysis was performed to report results by disease state.
Measure: Mean (Standard Deviation); unit: Percentage of red blood cells in blood
Arm/Group | Vadadustat
Number analyzed (Participants) | 10
Percentage of red blood cells in blood
  Baseline | 30.43 (2.69)
  Change from Baseline on Day 29 | 1.62 (1.71)
Statistical Analysis 1: Comparison: Vadadustat; Analysis of change from baseline on Day 29; Test type: Other — The test was based on Wilcoxon signed rank test, with an alpha level of 0.05; p = 0.0156, Wilcoxon signed rank test

3. Secondary Outcome: Mean Change From Baseline in Total Red Blood Cell (RBC) Count on Day 29
Description: Blood samples were collected to assess RBC count. Baseline RBC count was defined as the average of the 2 samples obtained prior to dosing (Pre-Baseline and Baseline). A positive change from baseline indicates RBC count increased.
Time Frame: Baseline; Day 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Million cells per cubic millimeter
Arm/Group | Vadadustat
Number analyzed (Participants) | 10
Million cells per cubic millimeter
  Baseline | 3.313 (0.389)
  Change from Baseline on Day 29 | 0.167 (0.170)
Statistical Analysis 1: Comparison: Vadadustat; Analysis of change from baseline on Day 29; Test type: Other — The test was based on Wilcoxon signed rank test, with an alpha level of 0.05; p = 0.0098, Wilcoxon signed rank test

4. Secondary Outcome: Mean Change From Baseline in Absolute Reticulocyte Count on Day 29
Description: Blood samples were collected to assess reticulocyte count. Baseline absolute reticulocyte count was defined as the average of the 3 reticulocyte counts obtained prior to dosing (Screening, Pre- Baseline, and Baseline). A positive change from baseline indicates absolute reticulocyte count increased.
Time Frame: Baseline; Day 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Cells per Microlitre
Arm/Group | Vadadustat
Number analyzed (Participants) | 10
Cells per Microlitre
  Baseline | 51076.00 (24975.76)
  Change from Baseline on Day 29 | 18647.00 (18289.84)
Statistical Analysis 1: Comparison: Vadadustat; Analysis of change from baseline on Day 29; Test type: Other — The test was based on Wilcoxon signed rank test, with an alpha level of 0.05; p = 0.0195, Wilcoxon signed rank test

5. Secondary Outcome: Mean Change From Baseline in Reticulocyte Hemoglobin (Hgb) Content on Day 29
Description: Blood samples were collected to assess reticulocyte Hgb. Baseline Hgb was defined as the average of the 2 samples obtained prior to dosing (Pre-Baseline and Baseline). A positive change from baseline indicates reticulocyte Hgb content increased.
Time Frame: Baseline; Day 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Vadadustat
Number analyzed (Participants) | 10
Picograms
  Baseline | 31.49 (2.44)
  Change from Baseline on Day 29 | 0.13 (0.84)
Statistical Analysis 1: Comparison: Vadadustat; Analysis of change from baseline on Day 29; Test type: Other — The test was based on Wilcoxon signed rank test, with an alpha level of 0.05; p = 0.8262, Wilcoxon signed rank test

6. Secondary Outcome: Number of Participants With Absolute Change From Baseline in Hemoglobin (Hgb) at Day 29
Description: Blood samples were collected to assess Hgb. Baseline Hgb was defined as the average of the 2 samples obtained prior to dosing (Pre-Baseline and Baseline).
Time Frame: Day 29
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vadadustat
Number analyzed (Participants) | 10
Participants
  Change from baseline ≥ 0.4 grams per decilitre | 6
  Change from baseline ≥ 0.6 grams per decilitre | 5
  Change from baseline ≥ 0.8 grams per decilitre | 3
  Change from baseline ≥ 1.0 grams per decilitre | 2

7. Secondary Outcome: Number of Participants With the Percentage Change From Baseline in Hemoglobin (Hgb) at Day 29
Description: as for outcome 6
Time Frame: Day 29
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vadadustat
Number analyzed (Participants) | 10
Participants
  Percent change from Baseline ≥ 5.0% | 5
  Percent change from Baseline ≥ 7.5% | 3
  Percent change from Baseline ≥ 10.0% | 3

8. Secondary Outcome: Number of Participants With Percentage Change From Baseline in Hematocrit at Day 29
Description: Blood samples were collected to assess hematocrit.
Time Frame: Day 29
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vadadustat
Number analyzed (Participants) | 10
Participants
  Percent change from Baseline ≥ 5.0% | 6
  Percent change from Baseline ≥ 7.5% | 2
  Percent change from Baseline ≥ 10.0% | 2

9. Secondary Outcome: Number of Participants With Percentage Change From Baseline in Red Blood Cell (RBC) Count at Day 29
Description: Blood samples were collected to assess RBC count. Baseline RBC count was defined as the average of the 2 samples obtained prior to dosing (Pre-Baseline and Baseline).
Time Frame: Day 29
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vadadustat
Number analyzed (Participants) | 10
Participants
  Percent change from Baseline ≥ 5.0% | 5
  Percent change from Baseline ≥ 7.5% | 3
  Percent change from Baseline ≥ 10.0% | 3

10. Secondary Outcome: Number of Participants With Change From Baseline in Absolute Reticulocyte Count at Day 29
Description: Blood samples were collected to assess reticulocyte count. Baseline absolute reticulocyte count was defined as the average of the 3 reticulocyte counts obtained prior to dosing (Screening, Pre- Baseline, and Baseline).
Time Frame: Day 29
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vadadustat
Number analyzed (Participants) | 10
Participants
  Change from Baseline ≥ 6000 cells per microlitre | 8
  Change from Baseline ≥ 12000 cells per microlitre | 7
  Change from Baseline ≥ 18000 cells per microlitre | 6

11. Secondary Outcome: Change From Baseline in Ferritin on Day 29
Description: Blood samples were collected to assess ferritin. A positive change from baseline indicates ferritin content increased.
Time Frame: Baseline; Day 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Nanograms per millilitre
Arm/Group | Vadadustat
Number analyzed (Participants) | 10
Nanograms per millilitre
  Baseline | 324.0 (199.2)
  Change from Baseline on Day 29 | -52.3 (36.6)
Statistical Analysis 1: Comparison: Vadadustat; Analysis of change from baseline on Day 29; Test type: Other — The test was based on Wilcoxon signed rank test, with an alpha level of 0.05; p = 0.0020, Wilcoxon signed rank test

12. Secondary Outcome: Change From Baseline in Iron on Day 29
Description: Blood samples were collected to assess iron. A positive change from baseline indicates iron content increased.
Time Frame: Baseline; Day 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Micrograms per decilitre
Arm/Group | Vadadustat
Number analyzed (Participants) | 10
Micrograms per decilitre
  Baseline | 69.4 (18.4)
  Change from Baseline on Day 29 | -8.2 (20.3)
Statistical Analysis 1: Comparison: Vadadustat; Analysis of change from baseline on Day 29; Test type: Other — The test was based on Wilcoxon signed rank test, with an alpha level of 0.05; p = 0.2383, Wilcoxon signed rank test

13. Secondary Outcome: Change From Baseline in Total Iron Binding Capacity on Day 29
Description: Blood samples were collected to assess total iron binding capacity. A positive change from baseline indicates total iron binding capacity increased.
Time Frame: Baseline; Day 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Micrograms per decilitre
Arm/Group | Vadadustat
Number analyzed (Participants) | 10
Micrograms per decilitre
  Baseline | 266.4 (56.4)
  Change from Baseline on Day 29 | 43.4 (34.8)
Statistical Analysis 1: Comparison: Vadadustat; Analysis of change from baseline on Day 29; Test type: Other — The test was based on Wilcoxon signed rank test, with an alpha level of 0.05; p = 0.0039, Wilcoxon signed rank test

14. Secondary Outcome: Change From Baseline in Transferrin Saturation on Day 29
Description: Blood samples were collected to assess transferrin saturation. The transferrin saturation is the ratio of the serum iron concentration and the total iron-binding capacity, expressed as a percentage. A positive change from baseline indicates transferrin saturation increased.
Time Frame: Baseline; Day 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Vadadustat
Number analyzed (Participants) | 10
Percentage
  Baseline | 26.1 (6.3)
  Change from Baseline on Day 29 | -6.4 (5.4)
Statistical Analysis 1: Comparison: Vadadustat; Analysis of change from baseline on Day 29; Test type: Other — The test was based on Wilcoxon signed rank test, with an alpha level of 0.05; p = 0.0039, Wilcoxon signed rank test

15. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An Adverse Event (AE) was defined as any untoward medical occurrence, signs, symptoms, disease, or laboratory or physiological observations occurring in a participant administered with drug, regardless of a causal relationship with that treatment or usage. This also included all suspected adverse medication reactions, reactions from medication overdose, abuse, withdrawal, sensitivity, toxicity, unrelated illnesses, including worsening a pre-existing condition, injury, or accidents. Serious Adverse Events (SAEs) was defined as any life-threatening condition; hospitalization or prolongation of existing hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect; or death.
Time Frame: Up to 2 weeks post 28 days of treatment
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vadadustat
Number analyzed (Participants) | 10
Participants
  TEAEs | 5
  SAEs | 0
  Deaths | 0

16. Secondary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Laboratory Parameter Values
Description: Parameters assessed for laboratory values included hematology, chemistry, urinalysis, and coagulation. The investigator was responsible for reviewing laboratory results for clinically significant changes.
Time Frame: Up to 2 weeks post 28 days of treatment
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vadadustat
Number analyzed (Participants) | 10
Participants | 0

17. Secondary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Vital Sign Values
Description: Parameters assessed for vital signs included sitting (at rest for a minimum of 5 minutes) heart rate, respiratory rate, body temperature, and blood pressure. The investigator was responsible for reviewing laboratory results for clinically significant changes.
Time Frame: Up to 2 weeks post 28 days of treatment
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vadadustat
Number analyzed (Participants) | 10
Participants | 0

18. Secondary Outcome: Number of Participants With Clinically Abnormal 12-Lead Electrocardiogram (ECG) Findings
Description: A standard 12-lead ECG was performed following dosing in a supine position for approximately 10 minutes. ECGs were taken prior to blood draws when possible. The investigator was responsible for reviewing laboratory results for clinical significance.
Time Frame: Up to 2 weeks post 28 days of treatment
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Vadadustat
Number analyzed (Participants) | 10
Participants | 0

19. Secondary Outcome: Mean Change From Baseline in PR Interval, QT Interval, QRS Interval, and QT Corrected (QTc) Interval
Description: A standard 12-lead ECG was performed following dosing in a supine position for approximately 10 minutes. ECGs were taken prior to blood draws when possible. The parameters evaluated from the participant ECG trace included PR interval, QT interval, QRS interval, and QTc (corrected).
Time Frame: Up to 2 weeks post 28 days of treatment
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Vadadustat
Number analyzed (Participants) | 10
Milliseconds
  Baseline PR Interval | 183.2 (42.6)
  Change from Baseline PR Interval | -4.4 (18.1)
  Baseline QT Interval | 415.6 (45.7)
  Change from Baseline QT Interval | 1.4 (20.3)
  Baseline QRS Interval | 95.4 (21.4)
  Change from Baseline QRS Interval | 3.4 (6.7)
  Baseline QTC Interval | 429.9 (30.5)
  Change from Baseline QTC Interval | 4.1 (8.3)

20. Secondary Outcome: Mean Trough Concentrations of Vadadustat at Day 8, 15, 22 and 29
Description: Serum samples were collected from the participants at the defined time points. Trough concentration was defined as the concentration of drug in the blood immediately before the next dose is administered. Trough concentration was calculated using the validated liquid chromatography-mass spectrometry (LC-MS) and liquid chromatography-tandem mass spectrometry (LC-MS/MS) method
Time Frame: Pre-dose at Day 8, 15, 22 and 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nanograms per millilitre
Arm/Group | Vadadustat
Number analyzed (Participants) | 10
nanograms per millilitre
  Day 8 | 3260.6 (2763.8)
  Day 15 | 3826.3 (2537.5)
  Day 22 | 3667.4 (1933.4)
  Day 29 | 5622.4 (5385.4)

ADVERSE EVENTS:
Time Frame: Up to 2 weeks post 28 days of treatment
Description: Treatment-emergent adverse events (TEAEs), defined as adverse events (AEs) that began (or pre-existing AEs that worsened) on or after the first dose through each participant's last participation date, were reported. Per the protocol, all results data are summarized as a single treatment arm (i.e., all participants receiving Vadadustat); no separate analysis was performed to report results by disease state.
Arm/Group | Vadadustat
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 5/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vadadustat (N=10)
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Chills (General disorders) | 1
Fatigue (General disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1

LIMITATIONS AND CAVEATS:
This pilot study planned to include 15 participants with either Stage 3 or 4 CKD, with no minimum or maximum enrollment target for either stage; however, because of slow enrollment the Sponsor terminated the study early after only 10 participants had enrolled. The overall status of the study was considered as completed since 10 participants received Vadadustat and all 10 participants completed the study per protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes